CLINICAL TRIAL: NCT01623947
Title: Effects of Sustamine(TM) on Cycling Time Trial Performance Following Prolonged Cycling
Brief Title: Effects of Sustamine(TM) on Cycling Time Trial Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Kyowa Hakko Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012-03-0043
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: glutamine; cycling performance; mental function

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Beverage
- 2.8 g Sustamine (Active Comparator)
  Interventions: Dietary Supplement: 2.8 g Sustamine Beverage
- 19.6 g Sustamine (Active Comparator)
  Interventions: Dietary Supplement: 19.6 g Sustamine Beverage

INTERVENTIONS:
Dietary Supplement: Placebo Beverage — 1400 ml flavored, colored, artificially sweetened, non-caloric beverage divided into 6 servings provided prior to and during the 2.5 hr interval ride.
  Arms: Placebo
Dietary Supplement: 2.8 g Sustamine Beverage — 1400 ml flavored, colored, artificially sweetened, beverage containing 2.8 g Sustamine divided into 6 servings provided prior to and during the 2.5 hr interval ride.
  Arms: 2.8 g Sustamine
Dietary Supplement: 19.6 g Sustamine Beverage — 1400 ml flavored, colored, artificially sweetened, beverage containing 19.6 g Sustamine divided into 6 servings provided prior to and during the 2.5 hr interval ride.
  Arms: 19.6 g Sustamine

SUMMARY:
Acute supplementation of Sustamine(TM), a combination of two amino acids, will improve cycling performance and mental acuity in a dose-dependent response.

ELIGIBILITY:
Inclusion Criteria:

* Competitive cyclist or triathlete
* Male (VO2max >= 55 ml/kg/min) or Female (VO2max >= 45 ml/kg/min)
* Healthy
* Blood pressure below 140/90
* Non-smoker

Exclusion Criteria:

* Anti-depressant medications
* Inconsistent regular medications
* Consumption performance-enhancing substances
* Type I or Type II diabetes
* Renal, hepatic or cardiac disease Current infectious disease

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Improved Time Trial Performance | After 2.5 hr interval cycling
  Participants will perform an interval ride on a cycling ergometer for 2.5 hr. Intervals will be at 50% or 75% of the participant's VO2max. The time trial will consist of 4 km up a constant grade.

SECONDARY OUTCOMES:
Improved Mental Function | After time trial
  Mental function will be assessed using a computer-based Stroop Test. Measurements will be collected before treatment, before exercise and after exercise.

CONTACTS AND LOCATIONS:
Overall Officials: John L. Ivy, Ph.D., Principal Investigator — University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States